CLINICAL TRIAL: NCT02422251
Title: Clinical Investigation of the Functional Outcomes of High Congruency Versus Low Congruency Knee Bearings
Brief Title: Biomechanical Assessment of a High Congruency Knee Bearing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: University of Strathclyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Ortho 14-12
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Knee Replacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mobile high congruency bearing (Experimental): Device B Braun Columbus total knee system using a rotating platform tibia and high congruency mobile bearing.
  Interventions: Device: Mobile high congruency bearing (Columbus)
- Fixed high congruency bearing (Experimental): Device B Braun Columbus total knee system using a fixed tibial platform and high congruency bearing.
  Interventions: Device: Fixed high congruency bearing (Columbus)
- Fixed low congruency bearing (Experimental): Device B Braun Columbus total knee system using a fixed tibial platform and low congruency bearing.
  Interventions: Device: Fixed high congruency bearing (Columbus)
- Control (No Intervention): Healthy control group

INTERVENTIONS:
Device: Mobile high congruency bearing (Columbus) — Columbus high congruency bearing on a rotating platform tibia.
  Arms: Mobile high congruency bearing
Device: Fixed high congruency bearing (Columbus) — Columbus high congruency bearing on a fixed platform tibia.
  Arms: Fixed high congruency bearing
Device: Fixed high congruency bearing (Columbus) — Columbus deep dish bearing on a fixed platform tibia.
  Arms: Fixed low congruency bearing

SUMMARY:
The aim of the project is to compare the biomechanics of three different bearing designs used in total knee replacement (TKR) implants. The bearing is the part in the middle of the knee implant that allows the metal tray attached to the shin bone (tibia) to move in relation to the metal part attached to the thigh bone (femur) and is usually made of plastic (high density polyethylene). There will be three different bearing types in the study, which all give different movements. This study will see which bearing is most like a natural knee and so which design gives the best function and feeling to patients with a TKR. 90 TKR patients from the Golden Jubilee National Hospital will be recruited and randomised to receive one of the three study bearings (30 in each group). In addition, a control group of 30 healthy individuals of similar age will be recruited for comparison. Before surgery and at 4 to 8 weeks and 1 year after their operation patients will attend biomechanical assessment sessions at the University of Strathclyde. The control group will attend the assessment session only once. In each of these sessions they will carry out a number of everyday tasks such as walking, moving from sitting to standing and going up and down stairs. These tasks will be measured using motion capture techniques. Reflective markers placed on each participant will be tracked by cameras so that their movements can be recorded. Force plates in the floor will record the forces during the tasks.

Movement and force data will be analysed to see if any differences exist between the groups and show which bearing gives the most natural movement.

DETAILED DESCRIPTION:
This is a double blind randomised controlled trial. The aim of the study is to compare the biomechanical performance of knee replacements with different bearing designs to that of a native or natural knee. The hypothesis is that a mobile bearing design with a high congruency bearing will allow the knee replacement to work more like the native knee and give more natural movement when carrying out everyday tasks.

The current evidence on whether fixed or mobile, low or high congruency bearings give the most natural movement or provide better knee function is sparse. By carrying out a randomised controlled trial including a cohort of healthy individuals and taking indepth functional assessments of a number of different common activities of daily living it should be possible to show what level of functional outcome the three bearings being used give.

Ninety patients scheduled for total knee arthroplasty under the care of four consultant orthopaedic surgeons at the Golden Jubilee National Hospital who meet the inclusion/exclusion criteria will be recruited and randomised into one of the three study groups (low congruency fixed bearing, high congruency fixed bearing or high congruency mobile bearing).

Invitation letters and participant information sheets will be sent out to suitable patients prior to their preoperative consultation. They will be approached at their consultation visit to seek consent to take part in the study. At this time they will be given the opportunity to ask questions about the study. Following written consent, the patient will be randomised using sequentially numbered opaque sealed envelopes. A nominated person, independent of the approach and consent of the patient, will sign and open the envelope and inform the hospital research team of the randomisation. The patient and the university research team will be blinded to randomisation. For each patient arrangements will be made for their preoperative movement analysis testing session. Subsequently, they will have their surgery and rehabilitation prior to discharge according to standard hospital practice. Participants will then return to the hospital for standard follow up appointments at six weeks and one year. At the same time arrangements will be made for them to attend their follow up movement analysis sessions. Clinical data recorded at preoperative assessment and postoperative follow up appointments, such as range of movement, Oxford Knee Score, patient satisfaction, EQ5D and radiographic measurements will be collected for study patients to compare to the functional outcomes measured during the movement analysis sessions.

Participants will be asked to attend movement analysis testing sessions at the University of Strathclyde in Glasgow on three separate occasions; preoperatively, at 4 to 8 weeks postoperatively and at one year postoperatively. Each of these sessions will follow the same procedure. Prior to data collection, participants will be asked to change into the tight fitting shorts and vest tops provided (male participants will be asked to forego the vest tops) in the changing rooms within the laboratory facility. Measurements of weight and body dimensions will be taken (required for processing the data) and then reflective markers will be attached to the legs, pelvis, torso and arms. These will be attached using toupee tape or elasticated straps as required. They will be asked to wear a headband (provided) with another four markers attached on their head. There will be eight activities of daily living (ADLs) in the test protocol, which will be carried out in one of two laboratories; one a standard motion capture laboratory (S) and the other in a laboratory with a CAREN system (Motek Medical, Amsterdam, Netherlands) which consists of a virtual reality screen, moving platform and treadmill (M). The ADLs will be:

1. Level walking in a straight line (S)
2. Level walking along a curved pathway (S)
3. Sit to stand to sit (S)
4. Sit to stand to walk (S)
5. Ascending and descending stairs (S)
6. Getting into and out of a car (S)
7. Single leg balance (M)
8. Walking on an incline (M)

Participants will be asked to perform each ADL in a fixed order several times until three good sets of data have been collected. Participants will be given instructions on how to perform each ADL prior to performing it and will be asked to practice them before data is collected. During the demanding tasks, participants will be supported by a harness to prevent falls and hand rails will be provided on the test staircase. Participants will be allowed rest breaks between each ADL and during tests if required. At the end of each task the participant will be asked a set of questions about how they found performing the task. On completion of the test protocol, the markers will be removed, the participant will get changed and will be free to leave. It is expected that each testing session will last up to 4 hours.

The three good data sets will be averaged to reduce variability. Statistical analysis will be carried out using an appropriate statistical package to determine if any significant differences exist in the data between the three patient groups and between the patient groups and the control group. All data will be tested for parametricity. Parametric data will be analysed using analysis of variance (ANOVA) tests with post hoc Bonferroni correction. If the data is found to be nonparametric, KruskalWallis tests will be used. For data over time appropriate repeated measures analysis will be used. A 95% confidence level will be used throughout.

The study is being funded over a three year period. The first year involves the set up and development of the protocol and the recruitment of the control participants. It is hoped that the recruitment of the patients will start nine months into the study period and will take 25 months to complete the data collection and analysis. This will allow two months for the reporting of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Primary unilateral total knee replacement
2. Suitable to have any one of the three test bearings
3. Over 35 years of age
4. Willing to take part
5. From one of the following NHS Scotland Health Boards: Ayrshire & Arran, Forth Valley, Greater Glasgow & Clyde, Highland, Lanarkshire or Lothian
6. Able to return for follow up sessions

Exclusion Criteria:

1. Previous hip or knee replacement procedure if carried out in the previous twelve months
2. Unable to give written consent
3. Unable to attend the movement analysis sessions
4. Journey time from home to the university in excess of two hours
5. Previous ankle surgery
6. Any past neurologic history e.g. stroke, Charcot-Marie-Tooth disease

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Knee kinematics | 1 year
  Knee range of motion during activities of daily living

SECONDARY OUTCOMES:
Hip kinematics | 1 year
  Hip range of motion during activities of daily living
Hip kinetics | 1 year
  Hip loading during activities of daily living
Knee kinetics | 1 year
  Knee loading during activities of daily living
Ankle kinematics | 1 year
  Ankle range of motion during activities of daily living
Ankle kinetics | 1 year
  Ankle loading during activities of daily living
EQ-5D | 1 year
  EQ-5D health questionnaire score
Oxford Knee Score | 1 year
  Oxford Knee Score questionnaire score
Knee alignment | 1 year
  Frontal plane alignment of the knee
Patient satisfaction | 1 year
  Score of patients' satisfaction with the implant
Complications | 1 year
  Evidence of any complication related to the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Picard, MD, Principal Investigator — National Waiting Times Centre
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

REFERENCES:
- [Derived] Komaris DS, Tedesco S, O'Flynn B, Govind C, Clarke J, Riches P. Dynamic stability during stair negotiation after total knee arthroplasty. Clin Biomech (Bristol). 2021 Jul;87:105410. doi: 10.1016/j.clinbiomech.2021.105410. Epub 2021 Jun 10. PMID 34130036
- [Derived] Komaris DS, Govind C, Murphy AJ, Clarke J, Ewen A, Leonard H, Riches P. Implant design affects walking and stair navigation after total knee arthroplasty: a double-blinded randomised controlled trial. J Orthop Surg Res. 2021 Mar 6;16(1):177. doi: 10.1186/s13018-021-02311-x. PMID 33676526